CLINICAL TRIAL: NCT04373564
Title: Prospective Evaluation of Potential Effects of Repeated Gadolinium-based Contrast Agent (GBCA) Administrations of the Same GBCA on Motor and Cognitive Functions in Neurologically Normal Adults in Comparison to a Non-GBCA Exposed Control Group
Brief Title: Effect on Body Movement and Mental Skills in Patients Who Received Gadolinium-based Contrast Media for Magnetic Resonance Examination Multiple Times Within 5 Years
Acronym: ODYSSEY
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Guerbet (Industry)
Collaborators: Bayer AG (Sponsor) (Unknown); Bracco (Sponsor) (Unknown); GEHC (Sponsor) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DGD-44-065; 20405 (Other: Bayer); GMRA-105 (Other: Bracco); GE-041-081 (Other: GE Healthcare); IQVIA-ODYS-001-LZA45541 (Other: IQVIA)
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Motor Function; Cognitive Function; Contrast Media
Keywords: Motor function assessment; Cognitive function assessment; Magnetic Resonance Imaging (MRI); Gadolinium; Gadolinium-based contrast agent (GBCA); Gadolinium retention; Breast cancer; Prostate cancer; Hepatocellular carcinoma; Colorectal cancer; Neuroendocrine tumor; Branch-duct intraductal papillary mucinous neoplasm (IPMN) of the pancreas
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Carcinoma, Hepatocellular; Colorectal Neoplasms; Neuroendocrine Tumors | interventions — Neuropsychological Tests; gadolinium ethoxybenzyl DTPA; gadobenic acid; gadodiamide; gadoterate meglumine; gadobutrol; gadoteridol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Linear GBCAs (Experimental): Adult participants, who were scheduled for repeated enhanced magnetic resonance imaging (MRI), receive a linear gadoliniumbased contrast agent (GBCA, i.e. Eovist/ Primovist, MultiHance or Omniscan) prior to MRI. Each participant will receive the same GBCA throughout the study.
  Interventions: Procedure: Motor Tests; Procedure: Cognitive Tests; Procedure: Unenhanced-MRI of the brain; Procedure: Gadolinium Measurements; Drug: Gadoxetate disodium; Drug: Gadobenate dimeglumine; Drug: Gadodiamide
- Macrocyclic GBCAs (Experimental): Adult participants, who were scheduled for repeated enhanced magnetic resonance imaging (MRI), receive a macrocyclic gadolinium-based contrast agent (GBCA, i.e. Gadavist/ Gadovist, Dotarem, Magnescope or ProHance) prior to MRI. Each participant will receive the same GBCA throughout the study.
  Interventions: Procedure: Motor Tests; Procedure: Cognitive Tests; Procedure: Unenhanced-MRI of the brain; Procedure: Gadolinium Measurements; Drug: Gadoterate meglumine; Drug: Gadobutrol; Drug: Gadoteridol
- No GBCA (Control arm) (Other): Adult participants who were never exposed to any gadolinium-based contrast agent and matching the population characteristics of the two GBCA arms. They will not receive any gadolinium-based contrast agent over the study course, but may undergo clinically indicated imaging (e.g. unenhanced magnetic resonance imaging (MRI), unenhanced or enhanced computed tomography, ultrasound and/or X-ray).
  Interventions: Procedure: Motor Tests; Procedure: Cognitive Tests; Procedure: Unenhanced-MRI of the brain; Procedure: Gadolinium Measurements

INTERVENTIONS:
Procedure: Motor Tests — To assess motor function annually
Procedure: Cognitive Tests — To assess cognitive function annually
Procedure: Unenhanced-MRI of the brain — The UE-MRI of the brain will be performed at baseline and at the year 5 visit in order to exclude presence of a significant MRI abnormality
Procedure: Gadolinium Measurements — Blood samples and spontaneous urine specimens will be collected through the course of the study to measure Gd concentration
Drug: Gadoxetate disodium — Administered as defined by the treating physician as part of routine clinical practice
  Other Names: Eovist; Primovist; BAY86-4873
  Arms: Linear GBCAs
Drug: Gadobenate dimeglumine — Administered as defined by the treating physician as part of routine clinical practice
  Other Names: MultiHance
  Arms: Linear GBCAs
Drug: Gadodiamide — Administered as defined by the treating physician as part of routine clinical practice
  Other Names: Omniscan
  Arms: Linear GBCAs
Drug: Gadoterate meglumine — Administered as defined by the treating physician as part of routine clinical practice
  Other Names: Dotarem; Magnescope
  Arms: Macrocyclic GBCAs
Drug: Gadobutrol — Administered as defined by the treating physician as part of routine clinical practice
  Other Names: BAY86-4875; Gadavist; Gadovist
  Arms: Macrocyclic GBCAs
Drug: Gadoteridol — Administered as defined by the treating physician as part of routine clinical practice
  Other Names: ProHance
  Arms: Macrocyclic GBCAs

SUMMARY:
This study is a postmarketing requirement jointly carried out by four NDA holders (Bayer AG, Bracco, GE Healthcare and Guerbet) and the CRO IQVIA.

The study aims to create detailed images of the organs and tissue of the human body during x-ray, CT-scan or MRI investigations, doctors are using contrast media (a kind of dye) which can be given to patients by injection into a blood vessel or by mouth.

In this study researchers want to find out whether so called gadolinium-based contrast agents (GBCAs) have an effect on body movement and mental skills when given to participants multiple times within 5 years.

The study plans to enroll about 2076 participants suffering from a condition for which they are likely to have at least annually a MRI or another imaging examinations. Only adults up to 65 years will be considered to join this study. During the study duration of 5 years participants will receive annually a MRI or other imaging tests (such as CT-scan, x-ray) and will visit the study doctor at least 7 times for physical examinations, laboratory investigations and tests on body movement and mental skills.

DETAILED DESCRIPTION:
The primary objective of the study is to assess the potential effect of repeated exposure to either a linear or a macrocyclic gadolinium-based contrast agent (GBCA) on change from baseline to Year 5 in composite measure of motor and cognitive function among neurologically normal adults in comparison to a matched non-GBCA- exposed control group.

The secondary objectives comprise the assessment of the following endpoints in GBCA-exposed participants as compared to controls a) changes from baseline in composite measure of motor and cognitive function post-baseline on yearly basis (Years 1 to 4); b) changes from baseline in each individual test of motor and cognitive function on yearly basis (Years 1 to 5). Total Gd concentrations in blood and urine samples on yearly basis (Years 1 to 5) and adverse events will be collected as secondary objectives.

Of note : The study is considered interventional because of the addition of UE-MRI scans for all participants, as well as blood sampling and the administration of the motor and cognitive tests. The GBCA administered as part of the contrast-enhanced MR imaging in the experimental arms is not the intervention in this study. Neither the protocol nor the investigators assign patients to a specific GBCA as part of the study, making this part of the study observational rather than interventional. The participants were already scheduled, prior to study screening, to undergo CE-MRI as part of their clinical care. The choice of GBCA for the CE-MRI will be based on medical need and institutional usage of GBCA, independent of study participation.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be neurologically normal, defined as free of unstable neurologic and psychiatric disease as confirmed by a normal neurologic examination at screening
* Participant (GBCA-exposed or controls) agrees to undergo unenhanced magnetic resonance imaging (UE-MRI) of the brain at enrollment and at the end of the observation period (5 years)
* Participants should have at least 1 of the following indications: a) Medium to high risk for breast cancer or dense breasts undergoing breast cancer screening with MRI, b) Elevated prostate-specific antigen (PSA) and under active diagnostic surveillance for prostate cancer, c) Chronic liver disease (eg, liver cirrhosis limited to Child class A, post-hepatitis chronic hepatopathy, or primary sclerosing cholangitis) for surveillance of hepatocellular carcinoma development, d) Low-grade colorectal cancer or neuroendocrine tumor undergoing screening for liver metastases or e) Branch-duct intraductal papillary mucinous neoplasm (IPMN) of the pancreas (maximum size ≤2 cm) undergoing imaging surveillance.

In addition, for participants in the GBCA Arms only:

* Each participant should be likely to undergo ≥5 GBCA-enhanced MR examinations with the same GBCA at least annually throughout the 5-year study duration
* Prospective participants with up to 3 well documented GBCA administrations prior to study screening are acceptable, provided that the imaging was performed with the same GBCA as the one to be prospectively used in the study. If the GBCA used cannot be identified, he/she cannot be enrolled.

For the Control Arm:

* Participants who never had and are not likely to receive any GBCA injection during the course of the study
* Each control participant must be willing to undergo UE-MRI of the brain at baseline and at Year 5. In Years 1 to 4, the control participants will undergo their clinically indicated UE-MRIs, computed tomography (CT), ultrasound, or X-ray procedures

Exclusion Criteria:

* As evidenced by history or determined in the neurologic exam at screening, concurrent neurological and/or psychiatric disease (or treatments) that could influence the results of the study's motor and cognitive tests (e.g. Cerebrovascular disease, Multiple sclerosis, Neurodegenerative disease, Malignant disease other than listed in indications, Carcinoid tumors, Epilepsy, Prior neurosurgery, Psychotic disorders or any prior psychotic episode not otherwise specified - any documented prior history of chronic schizophrenia, Remittent or current medically confirmed major depressive disorder or bipolar disorder, History of long-term major depression or bipolar affective disorder with an active episode in the past 2 to 5 years, Neurodevelopmental disorders (eg, trisomy 21), Uncontrolled severe migraine, Uncontrolled or controlled anxiety or depression within 6 months before enrollment, Screening scores of ≤24 on the MMSE and/or ≥11 on the Hospital Anxiety and Depression Scale (HADS)).
* Prior, planned, or ongoing chemotherapy or brain irradiation
* Use of concomitant medication(s) affecting neuro-cognitive or motor function
* Substance or alcohol abuse as determined by the investigator
* Alcoholic cirrhosis
* Renal disease, defined as estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2
* History of environmental/occupational/other exposure to one or more chemicals that may affect cognitive and/or motor function, including, but not limited to, heavy metals (arsenic [As], cadmium [Cd], lead [Pb], manganese [Mn], and mercury [Hg]), pesticides, solvents, or carbon monoxide.
* Clinical indications requiring >1 contrast enhanced magnetic resonance imaging (CE-MRI) every 6 months
* Pregnant or nursing (lactating) women
* Presence of any metal-containing joint implants/prostheses

In addition, for participants in either of the GBCA Arms only:

- Receipt of a GBCA or generic prior to study entry other than the specific GBCA to be administered during the course of the study.

For participants in the Control Arm only:

* Participants with any previous exposure to a GBCA.
* Participants with any contraindication to UE-MRI examinations.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2076 (Estimated)
Dates: Start 2021-03-24 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of motor function from baseline to year 5 in comparison to a matched non-GBCA-exposed control group | At baseline, year 5
  The endpoint is a composite z score, defined as the weighted sum of the z scores of the individual tests
Change in cognitive function from baseline to year 5 in comparison to a matched non-GBCA-exposed control group | At baseline, year 5
  The endpoint is a composite z score, defined as the weighted sum of the z scores of the individual tests

SECONDARY OUTCOMES:
Change from baseline in the composite endpoints (motor and cognitive) at each of the post-baseline time points (Years 1 to 4) in GBCA-exposed participants as compared to controls. | At baseline, years 1, 2, 3, 4
  The endpoint is a composite z score, defined as the weighted sum of the z scores of the individual tests
Change from baseline for each of the individual tests (motor and cognitive) at each of the post-baseline time points (Years 1 to 5) in GBCA-exposed participants as compared to controls. | At baseline, years 1, 2, 3, 4
  The endpoint is a composite z score, defined as the weighted sum of the z scores of the individual tests
Number of participants with adverse events | At baseline, years 1, 2, 3, 4, 5
Total Gd concentrations (as measured in a central laboratory) in blood and urine samples taken from exposed and control participants at the time of the annual visit | At baseline, years 1, 2, 3, 4, 5

CONTACTS AND LOCATIONS:
Locations (51):
- United States (16):
  - Scottsdale Medical Imaging, LLC, Scottsdale, Arizona
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Chicago Medical Center, Chicago, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Massachussets General Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - ActivMed Practices & Research, Inc., Methuen, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Department of Radiology, St Louis, Missouri
  - UNC School of Medicine, Chapel Hill, North Carolina
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Albert Einstein Healthcare Network, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin
- Brazil (10):
  - Hospital Santa Marta, Taguatinga, Federal District
  - Liga Norte-Rio-Grandense Contra o Câncer, Natal, Rio Grande do Norte
  - Instituto Mederi de Pesquisa e Saude, Passo Fundo, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Instituto Baía Sul de Ensino e Pesquisa (IEP), Florianópolis, Santa Catarina
  - CEMEC - Oncológica, São Bernardo do Campo, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - CPCLIN - Centro de Pesquisas Clínicas Ltda., São Paulo, São Paulo
  - Albert Einstein Sociedade Beneficente Israelita Brasileira, São Paulo, São Paulo
  - CEMEC - Oncológica, São Bernardo do Campo
- G. Kenneth Jansz Medical Professional Corporation, Burlington, Ontario, Canada
- France (2):
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - CHU Strasbourg - Hôpital Hautepierre, Strasbourg
- Germany (2):
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Vivantes Klinikum Neukoelln, Berlin
- Italy (5):
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena, Siena
  - Azienda Ospedaliera Universitaria di Trieste, Trieste, Trieste
  - Ospedale San Raffaele, Milan
  - Università Campus Bio-Medico di Roma, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona (Ospedale Borgo Roma), Verona
- Russia (7):
  - BHI of Omsk region "Clinical Oncology Dispensary", Omsk
  - FSBI "National medical scientific center of psychiatry and neurology n.a. V.M. Bekhterev" Adolescent, Saint Petersburg
  - FSBI North-West Federal Medical Research Center n.a. V.A. Almazov of MoH RF, Saint Petersburg
  - LLC Medical Center Mart, Saint Petersburg
  - RSBIH "Smolensk Regional Clinical Hospital", Smolensk
  - Federal State Budgetary Scientific Institution "Tomsk National Research Medical Centre of the Russia, Tomsk
  - SBIH Republican Clinical Oncological Dispensary of the MoH of Republic Bashkortostan, Ufa
- South Korea (8):
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do
  - Chonnam National University Hospital, Gwangju, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Inje University Busan Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Chosun University Hospital, Gwangju
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Chung-Ang University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No